CLINICAL TRIAL: NCT00192283
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled, Trial to Determine the Safety and Efficacy of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold-Adapted (CAIV-T) in Healthy Children Attending Day Care Centers
Brief Title: Trial to Determine the Safety and Efficacy of Influenza Virus Vaccine, Trivalent, Types A & B, Live Cold- Adapted (CAIV-T) in Healthy Children Attending Day Care Centers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Robert Walker, M.D., MedImmune Inc.
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: D153 P502
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluMist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): CAIV-T
  Interventions: Biological: CAIV-T
- 2 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: CAIV-T — The total single-dose volume of 0.2 mL was administered intranasally with the spray applicator intended for commercial use (approximately 0.1 mL into each nostril).
  Arms: 1
Other: Placebo — A single dose of placebo volume of 0.2 mL was administered intranasally with the spray applicator intended for commercial use (approximately 0.1 mL into each nostril).
  Arms: 2

SUMMARY:
The purpose of this study is to determine the efficacy of the liquid formulation of CAIVT against culture confirmed influenza illness in healthy children aged at least 6 months and less than 36 months, attending day care centers in Europe. In addition, the trial provides the opportunity to investigate the effect of CAIV-T on acute otitis media, on healthcare resource utilization and economic resources.

ELIGIBILITY:
Inclusion Criteria:

* who are aged at least 6 months and less than 36 months of age at the time of enrollment, attending day care for at least three days a week, four hours a day;
* who are in good health as determined by medical history, physical examination and clinical judgement;
* whose parent(s)/legal guardian(s) have provided written informed consent after the nature of the study has been explained;
* who, along with their parent(s)/legal guardian(s), will be available for duration of the trial (8 months ± 1 month);
* whose parent(s)/legal guardian(s), can be reached by study staff for the post-vaccination contacts [telephone, clinic or home visit].

Exclusion Criteria:

* whose parent(s)/legal guardian(s) are perceived to be unavailable or difficult to contact for evaluation or study visits during the study period;
* with any serious chronic disease (e.g., with signs of cardiac or renal failure or severe malnutrition), including progressive neurological disease;
* with Down's syndrome or other known cytogenetic disorders;
* with a known or suspected disease of the immune system or those receiving immunosuppressive therapy, including systemic corticosteroids; who received any blood products, including immunoglobulin, in the period from six months prior to vaccination through to the conclusion of the study;
* for whom there is intent to administer any other investigational vaccine or agent from one month prior to enrollment through to the conclusion of the study;
* have an immunosuppressed or an immunocompromised individual living in the same household; who, at any time prior to entry into this study, received a dose of any influenza vaccine (commercial or investigational);
* who, in the two weeks prior to entry into this study, received a dose of any influenza treatment (commercial or investigational);
* with a documented history of hypersensitivity to egg or egg protein or any other component of the study vaccine or placebo;
* with a clinically confirmed respiratory illness with wheezing within two weeks prior to enrollment;
* who received aspirin (acetylsalicylic acid) or aspirin-containing products in the two weeks prior to enrollment or for which use is anticipated during the study;
* who were administered any live virus vaccine within one month prior to enrollment or expected to receive another live virus vaccine within one month of vaccination in this study;
* with any medical conditions that in the opinion of the investigator might interfere with interpretation of the study results; If any of these criteria are met following enrolment, the subject will be excluded from subsequent vaccine dosing.

Note: A pregnant household member is not considered a contraindication to enrollment.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2903 (Actual)
Dates: Start 2000-09; Primary Completion 2002-04 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for efficacy is the first episode in a study child of a cultureconfirmed influenza illness. | 28 days after vaccination

SECONDARY OUTCOMES:
The secondary endpoint for culture-confirmed influenza illness is the first episode caused by any community-acquired antigenic subtype which occurs following receipt of the second dose of study vaccine or placebo. | 28 days after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walker, MD, Study Director — MedImmune LLC
Locations (1):
- Tampere University Medical School, Tampere, Finland